CLINICAL TRIAL: NCT05011032
Title: Effects of Homocysteine in Myocardial Infarction Patients in a Tertiary Care Hospital of Twin Cities of Pakistan
Brief Title: Effects of Homocysteine in Myocardial Infarction Patients in a Tertiary Care Hospital of Pakistan
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethical approval was not done. Hence the funding was withhold.
Sponsor: Aqua Medical Services (Pvt) Ltd (Industry)
Responsible Party: Principal Investigator, Mir Arif Hussain, Director, Aqua Medical Services (Pvt) Ltd
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Mubin 0011
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Homocystine; Metabolic Disorder
Keywords: Blood Sedimentation; Cardiovascular Diseases; Diabetes Mellitus; Homocysteine; Leukocytes; Cholesterol
MeSH Terms: conditions — Metabolic Diseases; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): The blood sample of 5ml was collected from the subjects via a sterile disposable 5ml syringe. The site for the blood collection was antecubital vein of the forearm, which was cleaned an alcoholic swab. The blood sample was shifted to assigned plain bottle container, where it was allowed to clot at room temperature. The serum sample was separated from the blood sample through a centrifugation process at a speed of 5000 revolutions per minute (rpm) for 15 minutes and stored frozen in another bottle container until the time for analysis
  Interventions: Diagnostic Test: Homocysteine
- Non-diabetic cardiac (Experimental): The blood sample of 5ml was collected from the subjects via a sterile disposable 5ml syringe. The site for the blood collection was antecubital vein of the forearm, which was cleaned an alcoholic swab. The blood sample was shifted to assigned plain bottle container, where it was allowed to clot at room temperature. The serum sample was separated from the blood sample through a centrifugation process at a speed of 5000 revolutions per minute (rpm) for 15 minutes and stored frozen in another bottle container until the time for analysis
  Interventions: Diagnostic Test: Homocysteine
- Diabetic cardiac (Experimental): The blood sample of 5ml was collected from the subjects via a sterile disposable 5ml syringe. The site for the blood collection was antecubital vein of the forearm, which was cleaned an alcoholic swab. The blood sample was shifted to assigned plain bottle container, where it was allowed to clot at room temperature. The serum sample was separated from the blood sample through a centrifugation process at a speed of 5000 revolutions per minute (rpm) for 15 minutes and stored frozen in another bottle container until the time for analysis
  Interventions: Diagnostic Test: Homocysteine

INTERVENTIONS:
Diagnostic Test: Homocysteine — It is an amino acid which is synthesized by the demethylation of dietary methionine. It is a highly reactive, Sulfur-containing amino acid as a by-product of metabolism of essential amino acid specifically methionine. It was proved to be a strong risk factor causing many cardiovascular diseases, neurological disturbances and other health related issues

SUMMARY:
Raised plasma Homocysteine (Hcy) was 1st proposed as a cause of vascular pathology in patients with inherited disorders of Homocysteine metabolism.leading to the hypothesis that individuals with slight to moderate elevated levels of Homocysteine may have an increased hazard for vascular disease. As an amino acid with a reactive sulfhydryl group, homocysteine has been proposed to intermediate vascular inflammation and damage by stimulating oxidative stress secondary to reactive oxygen species accumulation. which in turn leads to an rise in cardiac and vascular disease risk by stimulating endothelial dysfunction, smooth muscle cell proliferation, and vascular calcification. Consistent with this hypothesis, hyperhomocysteinemia a has been associated with an increased risk for coronary heart disease (CHD), heart failure, atrial fibrillation, stroke, and mortality.

DETAILED DESCRIPTION:
Excess of low density lipoproteins, high blood pressure, obesity, excess of blood sugar levels, smoking and sedentary life style are the known modifiable risk factors causing cardiovascular disease specifically Coronary disease. There can be some other substances which can additionally affect the human cardiac physiology as well i.e. high levels of Homocysteine molecule in the blood. The adverse effects of this component on multiple system of human body are evidenced in the literature since 1962 involving Nervous system, brain, Renal system, Liver functioning, Venus system and endothelial system and are still under debate. This biochemical agent has a strong relevance with the physiology of cardiovascular system and causes disturbance in the arterial supply of the heart in young population.

Homocysteine has been under a lot of discussion it is an amino acid which is synthesized by the demethylation of dietary methionine. It is a highly reactive, Sulfur-containing amino acid as a by-product of metabolism of essential amino acid specifically methionine. It was proved to be a strong risk factor causing many cardiovascular diseases, neurological disturbances and other health related issues. Homocysteine has a strong relation with the diseases involving hardening of arteries and blood clots related vascular problems.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years.
* Enough ability to complete the blood sampling procedure.
* Residents lived in the community and can walk to hospital.

Exclusion Criteria:

* Participants outside the age range.
* History of malignancy, infection and other comorbidities

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2021-09-09 (Estimated); Study Completion 2021-09-12 (Estimated)

PRIMARY OUTCOMES:
Homocysteine | 4th weeks
  It a marker of cardiovascular diseases.
Erythrocyte sedimentation rate (ESR) | 4th weeks
  It a marker of cardiovascular diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Mubin Kiyani, PhD, Principal Investigator — Shifa Tameer-e-Millat University
Locations (1):
- Mubin Kiyani, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karger AB, Steffen BT, Nomura SO, Guan W, Garg PK, Szklo M, Budoff MJ, Tsai MY. Association Between Homocysteine and Vascular Calcification Incidence, Prevalence, and Progression in the MESA Cohort. J Am Heart Assoc. 2020 Feb 4;9(3):e013934. doi: 10.1161/JAHA.119.013934. Epub 2020 Jan 30. PMID 32013703
- [Background] Balint B, Jepchumba VK, Gueant JL, Gueant-Rodriguez RM. Mechanisms of homocysteine-induced damage to the endothelial, medial and adventitial layers of the arterial wall. Biochimie. 2020 Jun;173:100-106. doi: 10.1016/j.biochi.2020.02.012. Epub 2020 Feb 24. PMID 32105811
- [Background] Sharma GS, Bhattacharya R, Singh LR. Functional inhibition of redox regulated heme proteins: A novel mechanism towards oxidative stress induced by homocysteine. Redox Biol. 2021 Oct;46:102080. doi: 10.1016/j.redox.2021.102080. Epub 2021 Jul 23. PMID 34325357
- [Background] Samarron SL, Miller JW, Cheung AT, Chen PC, Lin X, Zwerdling T, Wun T, Green R. Homocysteine is associated with severity of microvasculopathy in sickle cell disease patients. Br J Haematol. 2020 Aug;190(3):450-457. doi: 10.1111/bjh.16618. Epub 2020 Apr 19. PMID 32307711
- [Background] Paganelli F, Mottola G, Fromonot J, Marlinge M, Deharo P, Guieu R, Ruf J. Hyperhomocysteinemia and Cardiovascular Disease: Is the Adenosinergic System the Missing Link? Int J Mol Sci. 2021 Feb 8;22(4):1690. doi: 10.3390/ijms22041690. PMID 33567540
- [Background] Rong H, Huang L, Jin N, Hong J, Hu J, Wang S, Xie Y, Pu J. Elevated Homocysteine Levels Associated with Atrial Fibrillation and Recurrent Atrial Fibrillation. Int Heart J. 2020;61(4):705-712. doi: 10.1536/ihj.20-099. PMID 32727999
- [Background] Walli-Attaei M, Joseph P, Rosengren A, Chow CK, Rangarajan S, Lear SA, AlHabib KF, Davletov K, Dans A, Lanas F, Yeates K, Poirier P, Teo KK, Bahonar A, Camilo F, Chifamba J, Diaz R, Didkowska JA, Irazola V, Ismail R, Kaur M, Khatib R, Liu X, Manczuk M, Miranda JJ, Oguz A, Perez-Mayorga M, Szuba A, Tsolekile LP, Prasad Varma R, Yusufali A, Yusuf R, Wei L, Anand SS, Yusuf S. Variations between women and men in risk factors, treatments, cardiovascular disease incidence, and death in 27 high-income, middle-income, and low-income countries (PURE): a prospective cohort study. Lancet. 2020 Jul 11;396(10244):97-109. doi: 10.1016/S0140-6736(20)30543-2. Epub 2020 May 20. PMID 32445693
- [Background] Djurovic Z, Jovanovic V, Obrenovic R, Djurovic B, Soldatovic I, Vranic A, Jakovljevic V, Djuric D, Zivkovic V. The importance of the blood levels of homocysteine, folate and vitamin B12 in patients with primary malignant brain tumors. J BUON. 2020 Nov-Dec;25(6):2600-2607. PMID 33455102